CLINICAL TRIAL: NCT02658786
Title: Cost Effective Non Invasive Diagnostic Modalities and Predictive Model for Development and Progression of Fibrosis Among Patients With Hepatitis B, Hepatitis C Infection or Non Alcoholic Fatty Liver Disease: A Hospital Based Retrospective Followed by Prospective Cohort Study
Brief Title: Cost Effective Non Invasive Diagnostic Modalities and Predictive Model for Development and Progression of Fibrosis Among Patients With Hepatitis B, Hepatitis C Infection or Non Alcoholic Fatty Liver Disease
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-cohort-001
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2017-12

CONDITIONS: HBV; NAFLD; HCV
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hepatitis B patients: Biopsy proven Hepatitis B virus infected cases will be followed for the period of 5 years
- Hepatitis C patients: Biopsy proven Hepatitis C virus infected cases will be followed for the period of 5 years
- Non Alcoholic Fatty liver Disease patients: Biopsy proven Non Alcoholic Fatty liver Disease patients cases will be followed for the period of 5 years

SUMMARY:
Chronic liver diseases of differing etiologies are among the leading causes of morbidity and mortality worldwide [1]. Chronic liver disease progresses through different pathological stages that vary from mild hepatic inflammation without fibrosis to advanced hepatic fibrosis and cirrhosis [2]. Assessment of the stage of liver disease is important for diagnosis, treatment, and follow-up both during treatment and after cessation of treatment. A liver biopsy is the oldest and most accurate method used to evaluate liver histology and the progression of chronic liver disease. Furthermore, different histological scoring systems have been developed and modified [3]. A liver biopsy is considered the gold standard for assessing liver histology [4]. During the pathological progression of liver fibrosis, excessive amounts of extracellular matrix build up; furthermore, serum levels of various biomarkers change, in addition to the appearance of new biomarkers in the serum during the different stages of fibrosis [2, 5]. Recently many noninvasive markers (NIMs) for assessing liver fibrosis have been developed, and they are frequently used in clinical practice. They have been validated in different studies, and some were found to be highly accurate in the assessment of liver fibrosis compared with liver biopsies [6-7], which have always been used as the standard reference method for evaluating the accuracy of noninvasive methods. There are limited studies documenting the cost effectiveness of non invasive markers over invasive technique.

Most people with chronic Hepatitis B or C are unaware of their infection, putting them at serious risk of developing cirrhosis or liver cancer which are life threatening. Similarly patients with non alcoholic fatty liver diseases are unaware about fibrosis in liver. About 20-50% of persistent infection ends up into fibrosis and finally cirrhosis. Invasive and non invasive diagnostic methods are widely used to detect the fibrosis. Clinicians use different drugs and combinations to treat HBV and HCV infections. However, there is scarcity of a longitudinal prospective study to assess the cost effectiveness of these diagnostic measures.

We planned to conduct a retrospective followed by prospective cohort study among all cases that underwent biopsy in ILBS or GB Pant Hospital since 2000 till Dec 2020 with HBV infection, HCV infection, or non alcoholic fatty liver disease. For retrospective cohort study, we will collect data from hospital information system for all patients with HBV infection, HCV infection, or non alcoholic fatty liver disease, who underwent biopsy during the period of 2000-Dec 2015. The new patients with HBV infection, HCV infection, or non alcoholic fatty liver disease who will undergo biopsy during the period Jan 2016- Dec 2020 will serve as a cohort for prospective design.

We will collect socio-demographic data, clinical data, family history, personal history, medical history, anthropometry, biochemical and radiological data from each patient. We will also be conducting a cost effective analysis for various non invasive markers against biopsy as a gold standard in predicting fibrosis, both for retrospective and prospective cohorts.

For prospective cohort study, after evaluation of baseline biopsy results, the cases with metavir fibrosis score (F0-3) will be followed for a period of 5 years to document incidence of development and progression of fibrosis.

No additional investigation or test will be asked to the patient for the study. We will also develop a predicting model for development and progression of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Patients who underwent liver biopsy with underlying etiology as HBV, HCV, NASH or cryptogenic or ALD (inpatient or outpatient)
* Metavir Fibrosis Score F0-3 for prospective study design

Exclusion Criteria:

* Not willing to participate in the study
* Patients with chronic liver disease of other

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cases with Hepatitis B or Hepatitis C infection and Cases with non alcoholic fatty liver disease attending OPD or admitted in ward at ILBS, New Delhi
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of development & progression of fibrosis will be calculated. | 5 years
  Unit development and progression of fibrosis per person year.

SECONDARY OUTCOMES:
A predictive model for development & progression of fibrosis | 5 years
  Predictive model will be developed utilizing multiple regression analysis.
Validation of Non invasive markers for development and progression of fibrosis | 5 years
  Non invasive markers like ALT; AST/ALT ratio; AST/platelet ratio (APRI); Forns index; FIB-4 score; The FibroQ test; NAFLD fibrosis score; Lok Index and LSM (TE) will be calculated and tested against biopsy findings using ROC analysis.
Cost effective analysis for non invasive markers | 5 years
  Cost effective analysis will be done utilizing direct cost

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ajeet Singh Bhadoria, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No